CLINICAL TRIAL: NCT04176276
Title: Association Between Urinary and Serum Levels of miRNA 192 and miRNA 25 and Glomerular Filtration and Albuminuria in Patients With and Without Type 2 Diabetes.
Brief Title: Determining Serum and Urinary Levels of miRNA 192 and miRNA 25 in Patients With and Without Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, University of Pisa
Other Study IDs: AS0004
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Kidney Disease; Type2 Diabetes
Keywords: DKD; miRNA-25; miRNA-192
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urine, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Type2 Diabetes: 200 patients with type 2 diabetes consecutively enrolled among those referring to our Diabetes outpatient clinic.
  Interventions: Other: no interventions required.
- Patients without Type2 Diabetes: 100 patients without diabetes among those referring to our outpatient clinic most of them affected by hypercholesterolemia, obesity or CV disease.
  Interventions: Other: no interventions required.

INTERVENTIONS:
Other: no interventions required. — The study does not require any interventions.

SUMMARY:
Diabetes kidney disease (DKD) is the leading cause of end stage renal disease (ESRD) in western countries and its incidence is worryingly increasing worldwide. Cardiovascular disease shows a continuous relationship with declining of renal function in type 2 diabetes patients. Moreover, there is a strong evidence of all-cause mortality risk excess even in patients with early stages kidney disease.

MicroRNA (miRNA) are small non-coding RNA molecules, containing 21-25 nucleotides, that modulate post-transcriptional gene expressions. In the past years many human miRNAs involved in the pathogenesis of renal disease have been discovered, such as miR-192, miR-194, miR-204 and miR-25. Among these, miR-192 and miR-25, are receiving greater attention while it seems that they play a role in glomerulosclerosis and renal fibrosis. However too few data are available in large publish trials among patients with renal impairment and the role of serum and urinary levels of miR-192 and miR-25 in people with preserved renal function remain unclear.

To evaluate the association between serum and urinary expression of miR-192 and miR-25 and renal function (according to different extent of renal impairment) in patients with or without type 2 diabetes.

DETAILED DESCRIPTION:
The day of the study patients undergo a routine clinical evaluation. Whole blood samples are collected from an antecubital vein to assess serum/plasma aliquots of 200 μl each (frozen at -80°C until required for quantitation) for evaluation of biochemical parameters (fasting glucose, HbA1c, lipid profile, serum creatinine, uric acid, electrolytes, liver function enzymes, albumin) and determination of serum miR-192 and miR-25.

Two urine samples will be also collected to assess aliquots of 200 μl each (frozen at -80°C until required for quantitation) for determination of albumin:creatinine ratio and urine expression of miR-192 and miR-25.

ELIGIBILITY:
Inclusion Criteria (Group 1, Diabetic patients):

* age ≥ 18 years and ≤ 75 years
* male or female patients with type 2 diabetes treated with life style modification only or any OAD or insulin
* BMI ≥ 20 e ≤ 40 Kg/m2
* patients able to consent

Exclusion Criteria (Group 1, Diabetic patients):

* personal history of current or previous cancer or chemotherapy in the past 5 years
* personal history of alcohol and/or drugs abuse in the previous 3 months
* pregnancy

Inclusion Criteria (Group 2, Non-diabetic patients):

* age ≥ 18 years and ≤ 75 years
* BMI ≥ 20 e ≤ 40 Kg/m2
* patients able to consent

Exclusion Criteria (Group 2, Non-diabetic patients):

* diagnosis of type 2 or type 1 diabetes
* personal history of current or previous cancer or chemotherapy in the past 5 years
* personal history of alcohol and/or drugs abuse in the previous 3 months
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consecutively enrolled 300 patients (200 patients with type 2 diabetes and 100 patients without diabetes) among those referring to the Departiment of Diabetes and Metabolic disease, Santa Chiara Hospital, Pisa.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Serum expression of miR-192 | Each patients will be assessed at baseline.
  Levels of miR-192 will be assessed on serum and will be related to glomerular filtration rate and presence or absence of albuminuria (expressed as albumine:creatinine ratio).
Serum expression of miR-25 | Each patients will be assessed at baseline.
  Levels of miR-25 will be assessed on serum and will be related to glomerular filtration rate and presence or absence of albuminuria (expressed as albumine:creatinine ratio).
Urine expression of miR-192 | Each patients will be assessed at baseline.
  Levels of miR-192 will be assessed on urine and will be related to glomerular filtration rate and presence or absence of albuminuria (expressed as albumine:creatinine ratio).
Urine expression of miR-25 | Each patients will be assessed at baseline.
  Levels of miR-25 will be assessed on urine and will be related to glomerular filtration rate and presence or absence of albuminuria (expressed as albumine:creatinine ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solini, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy